CLINICAL TRIAL: NCT01960985
Title: Efficiency of Motor Training Program Associated With Extrenal Cues on the Balance of Patients With Parkinson's Disease.
Brief Title: Balance Training in Parkinson's Disease Using Cues
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tamine Capato 01
Record Dates: First submitted 2013-08-30; First posted 2013-10-11 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2013-10

CONDITIONS: Disturbance; Balance, Labyrinth; Parkinson´s Disease
Keywords: Balance, Postural; Parkinson´s Disease; H&Y 1-3; Exrecice; Postural adjustments; antecipatory postural; compensatory postural adjustments
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physicaltherapy (Experimental): Exprerimental group I - motor training balance training Exprerimental group II - motor training associated with visual and auditory cues on the balance training Control group - recived general orientations.
  Interventions: Other: Physicaltherapy
- physiotherapy (Experimental): Exprerimental group I - motor training balance training Exprerimental group II - motor training associated with visual and auditory cues on the balance training Control group - recived general orientations.
  Interventions: Other: Physicaltherapy

INTERVENTIONS:
Other: Physicaltherapy
  Other Names: balance training

SUMMARY:
Verifying the efficiency of motor training associated with visual and auditory cues on the balance, and postural anticipatory and compensatory adjustments of patients with Parkinson's Disease (PD), for prevent fall rate in people with PD. It is a single blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University.

DETAILED DESCRIPTION:
The objective of this work is verifying the efficiency of motor training associated with visual and auditory cues on the balance, and postural anticipatory and compensatory adjustments of patients with Parkinson's Disease (PD), for prevent fall rate in people with PD. It is a double blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University.

Forty two patients with idiopathic PD will take part in this study, at stages 2 to 3 of the Hoehn and Yahr Classification (HY). They are randomly assigned into one of 3 groups: one group receiving motor training associated to external cues (ET), the other one group performing motor training only (MT) and a third group receiving no treatment just generalize orientations. Performance in gait and balance are assessement before and after 10 training sessions (two 45-minute sessions per week) for the ET and MT groups, and before and after 5 weeks for the CG, using the BERG test (BT), Postural Stress Test (PST), Time Up and Go (TUG). Patients are also assessment for independence in daily life activities and motor performance using section II and III of the Unified Parkinson's Disease Rating Scale (UPDRS); for Quality of Life using the Parkinson's Disease Quality of Life (PDQL), and for emotional state by Beck's Depression Inventory (BDI). The training consist on: the experimental group receiving the motor program to balance associated to rhythmical auditory cues. The directions of the training were I. self-perception (strategies - Verbal and visual guidance); II. motor performance (Speed variation, Range of motion, Trunk mobility, Turning, balance exercices); III. Attention Strategies (Division of attention between guidance, environment and yourself movement, Maintenance of attention during all sets); IV. Cues.

The training program consisted on 5 weeks with 45 minutes duration, divided in 05 minutes warm-up, 30 minutes main part, 10 minutes cool down. The control group (CG) wasn't training just received orientations. Each session will consist on 05 minutes Warm-Up including: Muscle stretching, joint movements, upper and lower global, movement slowly and using wide joint movement range, and turning. The Main Part including: Head movement (bending, rotation, and leaning sideways), Axial and proximal movements, coordinated movements with Upper and Lower range and speed, Functional reach, weight shifts, stationary and walking gait with rhythmic and speed variation, postural reactions, trunk rotation, Balance exercises. And the last part is the Cool Down, including: Slow walk, breathing exercises associated to Upper limb movements and global muscular relaxation and stretching.

During the study there aren't changes on patient's usual medicine. The subjects will be reassessment after 4 and 30 weeks without the program training.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly
2. The patient is able to provide informed consent.
3. Definitive Idiopathic Parkinson's Disease as diagnosed by a Neurologist
4. Hoehn and Yahr Stage 1-3
5. Able to ambulate without an assistive device
6. On stable doses of Parkinson's medications prior to study onset

Exclusion Criteria:

1. Mini Mental Status Exam (MMSE) < 24
2. Change in Parkinson's medications in the duration of study
3. Uncontrolled orthostasis
4. Symptomatic coronary artery disease
5. Fracture of lower limb prior to study onset
6. Other neurologic diagnosis
7. Physical therapy before and during to study duration
8. Significant camptocormia
9. Any medical condition which the physician investigator determines would compromise the safety of exercise program for the subject.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
UPDRS | up to 30 weeks
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a rating scale used to follow the longitudinal course of Parkinson's disease

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) Berg Balance Scale | up to 30 weeks
  Berg Balance Scale assesses the functional balance of patients with Parkinson´s disease. It is a clinic assessment of patient that evaluate the antecipatory postural adjustments and the performance of patient to stand up and sit down, turn on and step, among others situations.
Dynamic Gait Index | up to 30 weeks
  The scale assesses the ability to adapt the gait during motor tasks with different demands
Retropulsion test | up to 30 weeks
  The Retropulsion test, by which an unexpected, quick and firm jerk on the shoulder is given in a backward direction.It is a clinic assessment of patient that evaluate the compensatory postural adjustments
Timed Up and Go test (TUG) | up to 30 weeks
  The Timed Up and Go test is a short, practical test by which gait and balance are tested
Balance Evaluation Systems Test (BESTest) | up to 30 weeks
  Clinical balance assessment tool that aims to target 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Tamine Capato, Master, Principal Investigator — University of Sao Paulo HCFMUSP; Maria Elisa Piemonte, PhG, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo Clinical Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886